CLINICAL TRIAL: NCT02739932
Title: Adolescent Mental Health: Canadian Psychiatric Risk and Outcome Study
Acronym: PROCAN
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Brain Canada (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Jean Addington, PhD, Professor, University of Calgary
Other Study IDs: MIRI-14-3377
Record Dates: First submitted 2016-03-22; First posted 2016-04-15 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder
Keywords: Attenuated Psychotic Symptoms
MeSH Terms: conditions — Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary study aims are to determine the clinical, behavioural and social predictors of SMI development in youth, and to investigate whether neuroimaging can distinguish youth who will develop SMI from those who will not.

The study's secondary aims are to examine the proportions of the cohort that make transitions between the different clinical stages of risk, and to determine the proportions that have poor outcomes, defined as ongoing or increased symptoms, secondary substance misuse, poor social or role functioning, i.e., non-participation in education, or employment, and new self-harm.

Investigators will study a cohort of 240 youth (aged 14-25, male and female) that includes youth with early mood symptoms or sub-threshold psychotic symptoms (symptomatic group; n=160), youth at risk due to a family history of a SMI (family high risk (FHR); n=40), and healthy controls (HC; n=40). From this cohort, clinical, social and cognitive data, as well as imaging data will be gathered to create a multi-layered "snapshot" of these individuals and provide full-level characterization. Investigators will use the full range of clinical and imaging data generated from this cohort to develop novel prediction algorithms incorporating key variables that predict the development of SMI.

ELIGIBILITY:
Inclusion Criteria:

* Participants will understand and sign an informed consent (or assent for minors) document in English.

Exclusion Criteria:

* meet criteria for current or lifetime Axis I bipolar or psychotic disorder (other Axis I disorders will not be exclusionary as they may be precursors to mood or psychotic disorders);
* IQ < 70;
* past or current history of a significant central nervous system disorder or serious medical disorder; and
* current pharmacological treatment that would be considered as an adequate trial of treatment for a SMI.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young people aged 12-25 who report 1 of the following:
  1. early mood symptoms or sub-threshold psychotic symptoms (n=160);
  2. a family history of a SMI (n=80); or
  3. are healthy with no mental health concerns (n=40).
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2015-03; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Diagnosis of serious mental illness (SMI) | 2 year
  The Structured Clinical Interview for DSM-IV Disorders (SCID-1) will be used to determine the presence of any Axis I disorder

SECONDARY OUTCOMES:
Level of risk on a Clinical Staging Model for Mental Health Disorders based on the Scale of Prodromal Symptoms (SOPS) | 2 year
  Level of risk will be defined based on a Clinical Staging Model for Mental Health Disorders (Hickie IB, Scott EM, Hermens DF et al. Applying clinical staging to young people who present for mental health care. Early Interv Psychiatry 2012.) Individuals will be assigned a stage based on their scores on the SOPS.
Level of risk on a Clinical Staging Model for Mental Health Disorders based on the Calgary Depression Scale for Schizophrenia (CDSS). | 2 year
  Level of risk will be defined based on a Clinical Staging Model for Mental Health Disorders (Hickie IB, Scott EM, Hermens DF et al. Applying clinical staging to young people who present for mental health care. Early Interv Psychiatry 2012.) Individuals will be assigned a stage based on scores on the CDSS.
Level of risk on a Clinical Staging Model for Mental Health Disorders based on the Young Mania Scale | 2 year
  Level of risk will be defined based on a Clinical Staging Model for Mental Health Disorders (Hickie IB, Scott EM, Hermens DF et al. Applying clinical staging to young people who present for mental health care. Early Interv Psychiatry 2012.) Individuals will be assigned a stage based on their scores on the Young Mania Scale.
Clinical symptoms on the Young Mania Scale. | 2 year
  Individuals' clinical symptoms will be measured using scores on the Young Mania Scale.
Clinical symptoms on the SOPS. | 2 year
  Individuals' clinical symptoms will be measured using scores on positive symptoms on the SOPS.
Clinical symptoms on the CDSS. | 2 year
  Individuals' clinical symptoms of depression will be measured using scores on the CDSS.
Functioning | 2 year
  Functioning will be assessed using Global Functioning (Social & Role)
Structural brain changes | 2 year
  MRI images will be examined for changes in structural data using regional grey matter intensity.
Structural Brain changes | 2 year
  MRI images will be examined for changes in structural data using white matter integrity
Functional Brain changes | 2 year
  MRI images will be examined for changes in functional data using resting-state connectivity among brain regions of interest
Changes in cognition | 2 year
  Cognition is assessed using the MATRICS Cognitive Battery

CONTACTS AND LOCATIONS:
Overall Officials: Jean Addington, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Mathison Centre for Research and Education, University of Calgary, Calgary, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario